CLINICAL TRIAL: NCT01839812
Title: Adrenal Responsiveness During the Perioperative Period in Children Undergoing Congenital Cardiac Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Sheri Crow, M.D., PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 08-001638
Record Dates: First submitted 2013-04-22; First posted 2013-04-25 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Adrenal Cortex Diseases; Infant Morbidity
Keywords: Cardiopulmonary bypass; Cortisol; Dexamethasone
MeSH Terms: conditions — Adrenal Cortex Diseases | interventions — Cosyntropin; Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cosyntropin stimulation test (Other): All patients enrolled in the study are administered cosyntropin stimulation tests to assess their adrenal response.
  Interventions: Drug: Cosyntropin

INTERVENTIONS:
Drug: Cosyntropin — A cosyntropin stimulation test is administered to each patient at 3 time points during the study to evaluate adrenal response.
  Other Names: adrenocorticotropic hormone

SUMMARY:
Our objective was to determine whether a standard 1mg/kg intraoperative dose of dexamethasone results in similar drug levels for all patients and to characterize the relationship between these drug levels and the innate stress response following infant Cardiopulmonary Bypass (CPB). The investigators hypothesized that postoperative dexamethasone levels are highly variable, and that the infant stress response is inversely related to the amount of dexamethasone measured in the blood. To test this theory the investigators simultaneously measured blood levels of dexamethasone and cortisol at critical time points during the perioperative period for infants undergoing CPB for CHD surgery.

DETAILED DESCRIPTION:
We conducted a single center prospective trial of infants (≤ 365 days of age) who presented to a single institution for congenital cardiac surgery.

Blood was collected from study participants at 7 time points; 1) post-anesthesia induction, 2) post-CPB/pre-MUF, 3) Intensive care unit (ICU) arrival, 4) post-op hour 4, 5) post-op hour 8, 6) post-op hour 12, and 7) post-op hour 24. At each of the 7 time points blood was analyzed for levels of the following; dexamethasone, cortisol, ACTH, Interleukin (IL) 10, IL 8, and IL 6. In addition, the innate stress response was evaluated with a cosyntropin stimulation test. Each patient received a 1 mcg/1.73 m2 intravenous dose of cosyntropin at; anesthesia induction, prior to dexamethasone (time 1), ICU arrival (time 3), and 24 hours after ICU arrival (time 7). Cortisol levels were measured before (time 1, 3, and 7) and 30 minutes after cosyntropin administration (time 1a, 3a, and 7a).

ELIGIBILITY:
Inclusion Criteria:

* less than 365 days of age
* Congenital cardiac surgery that requires cardiopulmonary bypass

Exclusion Criteria:

* Corticosteroids within 24 hours prior to enrollment
* Less than 36 weeks gestational age at time of surgery
* pre-operative mechanical circulatory support (ECMO)

Max Age: 365 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2009-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Cortisol level | 24 hours after surgery
  Primary outcome measure is the cortisol level for each patient at 7 time points throughout the operation and first 24 post-operative hours. Dexamethasone level of the patient is compared with the cortisol level.

CONTACTS AND LOCATIONS:
Overall Officials: Sheri S Crow, MD,MS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States